CLINICAL TRIAL: NCT07201610
Title: Non-invasive Diagnosis of Parkinson's Disease Using Hyperspectral Retinal Imaging, Optical Coherence Tomography, Computerized Cognitive Testing, and Voice Analysis
Brief Title: Non-invasive Diagnosis of Parkinson's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Blekinge Institute of Technology (Other)
Collaborators: Region Blekinge (Unknown)
Responsible Party: Sponsor
Other Study IDs: ps_hsi
Record Dates: First submitted 2025-09-12; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Parkinsons Disease (PD)
Keywords: Parkinson's disease; Non-invasive diagnosis; Hyperspectral retinal imaging; Optical coherence tomography; OCT; Computerized cognitive testing; Voice analysis; Biomarkers; Lewy body disease; Retinal biomarkers; Diagnostic accuracy; Neuropsychology; Machine learning
MeSH Terms: conditions — Parkinson Disease; Lewy Body Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson disease: Inclusion criteria for Parkinson's group:
  * Age 60-80 years
  * Diagnosis of idiopathic Parkinson's disease
  * Ability to understand spoken and written Swedish
  * Ability to personally provide consent to participate in the study
  * At least one healthy eye for retinal photography
- Healthy controls: Inclusion criteria for control group:
  * Age 60-80 years
  * Ability to understand spoken and written Swedish
  * Ability to personally provide consent to participate in the study
  * At least one healthy eye for retinal photography
  Definition of healthy:
  * No diagnosed Parkinson's disease or currently under investigation for Parkinson's disease
  * No diagnosed cognitive disease or currently under investigation for cognitive disease
  * No psychiatric disease affecting cognition (e.g., psychotic disorder or major depression)
  * Cognitive testing score of MMSE ≥ 26 points (out of a maximum of 30) and ≥ 8 points on the clock-drawing test

SUMMARY:
This study will investigate new, non-invasive methods to help diagnose Parkinson's disease. Researchers will use advanced eye imaging (hyperspectral retinal photography and OCT), computerized memory and thinking tests, and voice analysis to identify patterns linked to Parkinson's. The goal is to improve early and accurate diagnosis of Parkinson's disease without the need for spinal taps or invasive tests.

DETAILED DESCRIPTION:
This study aims to improve how Parkinson's disease is diagnosed by testing new, non-invasive techniques that do not require spinal taps or other invasive procedures. Researchers are investigating whether changes in the eye's retina, detected with hyperspectral imaging and optical coherence tomography (OCT), can help pinpoint Parkinson's disease. These methods use special photographs and scans, similar to those performed at an eye clinic or optometrist, to analyze patterns linked to nerve cells and blood vessels in the retina.

Additionally, participants will take computerized tests to measure memory, attention, and thinking skills. Since Parkinson's disease can also affect speech, the study will analyze voice recordings for specific changes that are common in the disease, such as reduced volume and strength. By combining information from eye images, cognitive tests, and voice analysis, the project hopes to develop a faster and more accurate way to diagnose Parkinson's disease at an earlier stage.

The study is open to both people with Parkinson's disease and healthy volunteers, and the new diagnostic tools being tested could make future diagnosis simpler, more comfortable, and accessible to a wider population

ELIGIBILITY:
Inclusion criteria for Parkinson's group:

* Age 60-80 years
* Diagnosis of idiopathic Parkinson's disease
* Ability to understand spoken and written Swedish
* Ability to personally provide consent to participate in the study
* At least one healthy eye for retinal photography

Inclusion criteria for control group:

* Age 60-80 years
* Ability to understand spoken and written Swedish
* Ability to personally provide consent to participate in the study
* At least one healthy eye for retinal photography
* Healthy as defined below

Exclusion criteria:

* At least one eye must not have retinal disease, glaucoma, or vascular eye disease (such as embolism)
* Angle-closure glaucoma or other contraindication to mydriatic drops
* Low functional ability that makes participation in examinations impossible
* Diagnosed dementia
* Specifically for the control group: Not healthy according to the definition below

Definition of healthy:

* No diagnosed or suspected Parkinson's disease
* No diagnosed or suspected cognitive disease
* No psychiatric disease affecting cognition (e.g., psychotic disorder or major depression)
* Cognitive testing with MMSE ≥ 26 points (out of a maximum of 30) and ≥ 8 points on the clock-drawing test

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thirty consecutive patients with a diagnosis of idiopathic Parkinson's disease who are scheduled for routine follow-up visits at the Neurology Clinic in Karlskrona.
  After patient recruitment, 30 healthy controls matched by age and gender (1:1 matching) will be recruited from Blekinge Institute of Technology's (BTH) Research and Development Clinic. At the clinic, there is a list/mailbox where individuals can volunteer to participate in studies. The participants who best match the included Parkinson's patients will be invited to take part
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10-16 (Estimated); Primary Completion 2025-12-16 (Estimated); Study Completion 2025-12-16 (Estimated)

PRIMARY OUTCOMES:
Performance of combined model, retinal, voice and cognitive data | Through study completion, an average of 6 months
  To assess the performance (AUC) of an optimized diagnostic model that combines HSI, OCT, and angio-OCT data with computerized cognitive testing and voice analysis for identifying Parkinson's disease
Performance retinal biomarkers | Through study completion, an average of 6 months
  To evaluate the performance (AUC) of a diagnostic model that combines hyperspectral retinal imaging (HSI), and optimally selected data from OCT and angio-OCT, for classifying patients with Parkinson's disease

SECONDARY OUTCOMES:
Diagnostic performance of each modality on its own. | Through study completion, an average of 6 months
  Diagnostic performance for each diagnostic modality, HSI, OCT, voice and cognitive testing
Correlational analyses | Through study completion, an average of 6 months
  Correlation measures for each retinal modality with cognition and functional scale for Parkinson's disease

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be shared upon request from a regarded trustworthy academic partner for replicating purposes only.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication
Access Criteria: Anonymised data will be shared upon request from a regarded trustworthy academic partner for replicating purposes only.